CLINICAL TRIAL: NCT01723735
Title: A Randomized, Partial Blind, 3 Parallel Groups Study of the Pharmacodynamic Profile of SAR236553 (REGN727) Administered as Multiple Subcutaneous Doses, Either Alone or on Top of Ezetimibe or Fenofibrate Administered as Multiple Oral Doses in Healthy Subjects
Brief Title: Effect of Alirocumab (SAR236553/REGN727) Administered on Top of Ezetimibe or Fenofibrate on Lipid Profiles in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PKD12910; U1111-1131-3203 (Other: UTN); 2012-003049-13 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Ezetimibe; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alirocumab + Ezetimibe Placebo (Experimental): Subcutaneous (SC) injections of alirocumab added to oral administration of ezetimibe placebo
  Interventions: Drug: Alirocumab; Drug: Ezetimibe Placebo
- Alirocumab + Ezetimibe (Experimental): Subcutaneous (SC) injections of alirocumab added to oral administration of ezetimibe
  Interventions: Drug: Alirocumab; Drug: Ezetimibe
- Alirocumab + Fenofibrate (Experimental): Subcutaneous (SC) injections of alirocumab added to oral administration of fenofibrate
  Interventions: Drug: Alirocumab; Drug: Fenofibrate

INTERVENTIONS:
Drug: Alirocumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: SAR236553; REGN727
Drug: Ezetimibe — Pharmaceutical form: overencapsulated tablet
  Route of administration: oral
  Arms: Alirocumab + Ezetimibe
Drug: Ezetimibe Placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: Alirocumab + Ezetimibe Placebo
Drug: Fenofibrate — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Alirocumab + Fenofibrate

SUMMARY:
Primary Objective:

To assess the pharmacodynamic profile of alirocumab (SAR236553/REGN727) administered either alone or on top of ezetimibe or fenofibrate, based on low-density lipoprotein -cholesterol (LDL-C).

Secondary Objectives:

* To assess the pharmacodynamic profile of alirocumab administered either alone or on top of ezetimibe or fenofibrate, based on other lipid parameters.
* To assess the pharmacokinetic profile of alirocumab administered either alone or on top of ezetimibe or fenofibrate.

DETAILED DESCRIPTION:
Total duration of the study per subject (excluding screening) is about 22 weeks.

ELIGIBILITY:
Inclusion criteria :

* Healthy male /or female subjects,
* aged 18 to 65 years old,
* with LDL-C > 130 mg/dL
* not receiving lipid lowering therapy.

Exclusion criteria:

* Healthy subjects with history or presence of clinically relevant illness.
* Subjects currently taking statins, ezetimibe or fenofibrate.
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of alirocumab on LDL-C | Up to 18 weeks

SECONDARY OUTCOMES:
Assessment of the pharmacodynamic profile of alirocumab | Up to 18 weeks
Pharmacokinetics: Assessment of serum concentrations of alirocumab | Up to 18 weeks
Pharmacokinetics: Assessment of serum concentrations of proprotein convertase subtilisin kexin type 9 (PCSK9) | Up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- France (2):
  - Investigational Site Number 250001, Rennes
  - Investigational Site Number 250002, Rueil-Malmaison

REFERENCES:
- [Result] Rey J, Poitiers F, Paehler T, Brunet A, DiCioccio AT, Cannon CP, Surks HK, Pinquier JL, Hanotin C, Sasiela WJ. Relationship Between Low-Density Lipoprotein Cholesterol, Free Proprotein Convertase Subtilisin/Kexin Type 9, and Alirocumab Levels After Different Lipid-Lowering Strategies. J Am Heart Assoc. 2016 Jun 10;5(6):e003323. doi: 10.1161/JAHA.116.003323. PMID 27287699